CLINICAL TRIAL: NCT03147703
Title: Timing of Food Intake Impacts Daily Rhythms of Human Saliva Microbiota in a Mediterranean Population
Brief Title: Timing of Food Intake Impacts Daily Rhythms of Human Saliva Microbiota
Acronym: ONTIME-MIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, PROF. MARTA GARAULET AZA, Full profesor, Universidad de Murcia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2017ES00003
Record Dates: First submitted 2017-04-25; First posted 2017-05-10 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Healthy Women
Keywords: Microbiota; Food timing; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Eating (EE) (Experimental): The intervention is Food Timing, Early Eating is defined at 13:00 hours for lunch
  Interventions: Behavioral: Food Timing
- Late Eating (LE) (Experimental): The intervention is Food Timing, Late Eating is defined for 17:30 hours for lunch
  Interventions: Behavioral: Food Timing

INTERVENTIONS:
Behavioral: Food Timing — the timing of the main meal of the day (lunch in Spain) is changed from early (14:00) to late (17:30) and viceversa in a randomized and crossover way

SUMMARY:
The purpose of this investigation is to test the hypothesis that in humans, eating late may induce changes in saliva microbiota daily rhythms towards a more obesogenic and a less responsiveness to dietary treatments profile. These changes in microbiota may partly explain the weight loss difficulties that characterized late eaters in previous studies. Thus, the aim is to analyze the effect of the timing of food intake in humans' saliva microbiome daily rhythms in a randomized, crossover interventional study, in order to achieve.

DETAILED DESCRIPTION:
Overweight and obesity can currently be considered a major threat to human health. Recent studies suggest that not only "what" we eat, but also "when" we eat may have a significant role in obesity treatment. The importance of caloric distribution across the day on weight loss therapy was supported by a 12-weeks experimental study showing that subjects assigned to high caloric intake during breakfast lost significantly more weight than those assigned to high caloric intake during the dinner. These results suggest that eating late may affect obesity and impair the success of weight loss therapies.

Novel evidence from animal and human studies indicates that the composition of the gut microbiota may also be involved in obesity and weight loss. Moreover, studies performed in extreme obese subjects have demonstrated that weight loss improves the obesity-associated gut microbiota composition towards a lean microbiome phenotype.

A recent study has shown that the timing of food intake influences microbiota in mice model. This study reported that obesity dampens the cyclical changes in the gut microbiome of mice while time-restricted feeding (TRF), in which feeding is consolidated to the nocturnal phase, partially restores these cyclical fluctuations. Furthermore, TRF which protects against obesity and metabolic diseases affects bacteria and has shown to influence host metabolism. Then, feeding pattern and time of food intake, in addition to diet, are important parameters when assessing the microbiome's contribution to mice metabolism. However, to our knowledge no human studies are available showing the effect of timing of food intake in microbiota.

Thus, the aim was to analyze the effect of the timing of food intake in humans' saliva microbiome, in order to achieve a better understanding of the relationship between food timing, obesity and weight loss in humans.

This goal will be achieved through a specific approach:

• Interventional (randomized, cross-over controlled trials) (Aim 1): To study that, eating late may induce changes in saliva microbiota daily rhythms towards a more obesogenic pattern and a less responsiveness to dietary treatments profile in women (n=10).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Body Mass Index: 20 to 30 kg/m2
* Caucasian
* Day workers

Exclusion Criteria:

* Endocrine (Diabetes mellitus or others), renal, hepatic, cancer or psychiatric disorders
* Receiving any pharmacologic treatment other than oral contraceptives
* Bulimia diagnosis, prone to binge eating
* Pregnancy

Ages: 20 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Saliva microbiome daily rhythms | Total of 4 weeks. Samples will be collected after week 1 and 2 and at week 4.
  Investigators will measure daily rhythms of saliva microbiome at early eating and late eating visits.
Feces microbiome daily rhythms | Total of 4 weeks. Samples will be collected after week 1 and 2 and at week 4.
  Investigators will assess gut microbiome with one feces sample at early eating and late eating visits.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Garaulet, PHD, Study Director — Universidad de Murcia
Locations (1):
- University of Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No
Spain: Ministry of Health and consumption